CLINICAL TRIAL: NCT02042963
Title: KoreaN Cohort Study for Outcome in Patients With Kidney Transplantation : A 9-year Longitudinal Cohort Study of the Kidney Transplantation (KNOW-KT)
Brief Title: KoreaN Cohort Study for Outcome in Patients With Kidney Transplantation (KNOW-KT)
Acronym: KNOW-KT
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Seoul National University Hospital (Other)
Collaborators: Asan Medical Center (Other); Chonbuk National University Medical School (Unknown); Gachon University Gil Medical Center (Other); Keimyung University Dongsan Medical Center (Other); Korea University (Other); Kyungpook National University Hospital (Other); Samsung Medical Center (Other); Medical Research Collaborating Center, Seoul, Korea (Other); Yonsei University (Other); Seoul National University College of Medicine (Unknown)
Responsible Party: Principal Investigator, Curie Ahn, Professor, Seoul National University Hospital
Other Study IDs: KNOW-KT
Record Dates: First submitted 2014-01-20; First posted 2014-01-23 (Estimated); Last update posted 2014-01-23 (Estimated); Status verified 2014-01

CONDITIONS: Kidney Transplant Recipients; Complications After Kidney Transplant
Keywords: The cohort of Asian kidney transplant recipients; The cohort of metabolic complication after kidney transplant; The biorepository of Asian kidney transplant recipients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Years
Biospecimen Retention: Samples With DNA — DNA, serum, urine, RNA (blood and urine)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- KNOW-KT: 1000 Kidney transplant recipients in Korea

SUMMARY:
KNOW-KT (KoreaN cohort study for Outcome in patients With KT: A 9-year Longitudinal cohort study of the Korean adult KT patients), funded by Korea Center for Disease Control and Prevention (KCDC) was established in 2012 by a group of transplant physicians, transplant surgeons, nephrologists, epidemiologists, and biostatisticians in Korea.

We aimed to establish an adult KT cohort, to investigate the renal allograft outcomes, mortality, complications, and to explore traditional or nontraditional risk factors for morbidity and mortality. We established a bio-bank to integrate clinical and biological information. Here, we report design and method of the KNOW-KT.

ELIGIBILITY:
Inclusion Criteria:

* Recipients and Donors of kidney transplant

Exclusion Criteria:

* Multi-organ transplant recipients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Kidney transplant recipients and their donors (donors for baseline data)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2012-03; Primary Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
overall mortality | 9 years
Allograft survival | 9 years
  defined as re-transplant or initiation of maintenance dialysis

SECONDARY OUTCOMES:
cardiovascular event | 9 years
  Acute Myocardial Infarction Revascularization : PCI or CABG Stroke Admission from Congestive heart failure
Albuminuria | 9 years
Acute Rejection | 9 years
New onset of diabetes after transplant | 9 years
Quality of Life | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National Univeristy Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Jung HY, Jeon Y, Huh KH, Park JB, Kim MG, Lee S, Han S, Ro H, Yang J, Ahn C, Cho JH, Park SH, Kim YL, Kim CD. Pretransplant and Posttransplant Alcohol Consumption and Outcomes in Kidney Transplantation: A Prospective Multicenter Cohort Study. Transpl Int. 2022 May 30;35:10243. doi: 10.3389/ti.2022.10243. eCollection 2022. PMID 35707634
- [Derived] Hong N, Lee J, Kim HW, Jeong JJ, Huh KH, Rhee Y. Machine Learning-Derived Integer-Based Score and Prediction of Tertiary Hyperparathyroidism among Kidney Transplant Recipients: An Integer-Based Score to Predict Tertiary Hyperparathyroidism. Clin J Am Soc Nephrol. 2022 Jul;17(7):1026-1035. doi: 10.2215/CJN.15921221. Epub 2022 Jun 10. PMID 35688469
- [Derived] Yang J, Lee J, Huh KH, Park JB, Cho JH, Lee S, Ro H, Han SY, Kim YH, Jeong JC, Park BJ, Han DJ, Park SB, Chung W, Park SK, Kim CD, Kim SJ, Kim YS, Ahn C; KNOW-KT Study Group. KNOW-KT (KoreaN cohort study for outcome in patients with kidney transplantation: a 9-year longitudinal cohort study): study rationale and methodology. BMC Nephrol. 2014 May 9;15:77. doi: 10.1186/1471-2369-15-77. PMID 24884405